CLINICAL TRIAL: NCT04312009
Title: Randomized Controlled Trial of Losartan for Patients With COVID-19 Requiring Hospitalization
Brief Title: Losartan for Patients With COVID-19 Requiring Hospitalization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SURG-2020-28675; INV-017069 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Corona Virus Infection; Acute Respiratory Distress Syndrome; SARS-CoV Infection
Keywords: COVID-19; Corona Virus; SARS-COV-2
MeSH Terms: conditions — Coronavirus Infections; Respiratory Distress Syndrome; Severe Acute Respiratory Syndrome; COVID-19 | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Losartan (Experimental): Participants in this arm will receive the study drug, Losartan.
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Losartan — Losartan; 50 mg daily; oral administration
  Other Names: Cozaar
  Arms: Losartan
Other: Placebo — Placebo (microcrystalline methylcellulose, gelatin capsule); oral administration
  Arms: Placebo

SUMMARY:
This is a multi-center, double-blinded study of COVID-19 infected patients requiring inpatient hospital admission randomized 1:1 to daily Losartan or placebo for 7 days or hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Presumptive positive laboratory test for Covid-19 based on local laboratory standard
* Age greater than or equal to 18 years of age
* Admission to the hospital with a respiratory SOFA >=1 and increased oxygen requirement compared to baseline among those on home O2
* Randomization within 48 hours of presentation of hospital admission or within 48 hours of a positive test result, whichever is later

Exclusion Criteria:

* Randomization > 48 hours of admission order or positive test result, whichever is later
* Currently taking an angiotensin converting enzyme inhibitor (ACEi) or Angiotensin receptor blocker (ARB)
* Prior reaction or intolerance to an ARB or ACE inhibitor, including but not limited to angioedema
* Pregnant or breastfeeding
* Lack of negative urine or serum pregnancy test
* Not currently taking a protocol allowed version of contraception: intrauterine device, Depo-formulation of hormonal contraception (e.g. medroxyprogesterone acetate / Depo-Provera), subcutaneous contraceptive (e.g. Nexplanon), daily oral contraceptives with verbalized commitment to taking daily throughout the study period; use of condoms or agree to abstain from sexual intercourse during the study. All women of child bearing age enrolled in this fashion will be informed of the teratogenic risks. If enrolled under LAR, they will be informed of the risks after regaining capacity.
* Patient reported history or electronic medical record history of kidney disease, defined as:

  1. Any history of dialysis
  2. History of chronic kidney disease stage IV
  3. Estimated Glomerular Filtration Rate (eGFR) of < 30ml/min/1.73 m2 at the time of randomization
* Severe dehydration at the time of enrollment in the opinion of the investigator or bedside clinician
* Most recent mean arterial blood pressure prior to enrollment <65 mmHg
* Patient reported history or electronic medical record history of severe liver disease, defined as:

  1. Cirrhosis
  2. History of hepatitis B or C
  3. Documented AST or ALT > 3 times the upper limit of normal measured within 24 hours prior to randomization
* Potassium >5.0 within 24 hours prior to randomization unless a repeat value was <=5.0
* Treatment with aliskiren
* Inability to obtain informed consent from participant or legally authorized representative
* Enrollment in another blinded randomized clinical trial for COVID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Tignanelli, MD, Principal Investigator — University of Minnesota; Michael Puskarich, MD, MS, Principal Investigator — University of Minnesota
Locations (13):
- United States (13):
  - University of Florida Health Gainesville, Gainesville, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - M Health Fairview Ridges Hospital, Burnsville, Minnesota
  - M Health Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - North Memorial Health Hospital, Robbinsdale, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cooper University Hospital, Camden, New Jersey
  - University of Cincinnati Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puskarich MA, Ingraham NE, Merck LH, Driver BE, Wacker DA, Black LP, Jones AE, Fletcher CV, South AM, Murray TA, Lewandowski C, Farhat J, Benoit JL, Biros MH, Cherabuddi K, Chipman JG, Schacker TW, Guirgis FW, Voelker HT, Koopmeiners JS, Tignanelli CJ; Angiotensin Receptor Blocker Based Lung Protective Strategies for Inpatients With COVID-19 (ALPS-IP) Investigators. Efficacy of Losartan in Hospitalized Patients With COVID-19-Induced Lung Injury: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e222735. doi: 10.1001/jamanetworkopen.2022.2735. PMID 35294537
- [Derived] Smolander J, Bruchfeld A. [COVID-19 and kidney disease]. Lakartidningen. 2020 Jul 13;117:20110. Swedish. PMID 32658300

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Losartan
Started | 104 | 101
Completed | 102 | 100
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Losartan | Total
Number analyzed (Participants) | 104 | 101 | 205
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 78 | 158
  >=65 years | 24 | 23 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 63 | 60 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 7 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 30 | 37 | 67
  White | 47 | 35 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Difference in Estimated (PEEP Adjusted) P/F Ratio at 7 Days
Description: Outcome calculated from the partial pressure of oxygen or peripheral saturation of oxygen by pulse oximetry divided by the fraction of inspired oxygen (PaO2 or SaO2 : FiO2 ratio). PaO2 is preferentially used if available. A correction is applied for endotracheal intubation and/or positive end-expiratory pressure. Patients discharged prior to day 7 will have a home pulse oximeter send home for measurement of the day 7 value, and will be adjusted for home O2 use, if applicable. Patients who died will be applied a penalty with a P/F ratio of 0.
Time Frame: 7 days
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 102 | 100
ratio | 281.4 [256.7 to 306.1] | 260.9 [234.1 to 287.8]

2. Secondary Outcome: Daily Hypotensive Episodes
Description: Outcome reported as the mean number of daily hypotensive episodes (MAP < 65 mmHg) prompting intervention (indicated by a fluid bolus >=500 mL) per participant in each arm.
Time Frame: 10 days
Measure: Mean (95% Confidence Interval); unit: episodes per day
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 102 | 100
episodes per day | 0.048 [0.018 to 0.1] | 0.119 [0.065 to 0.191]

3. Secondary Outcome: Proportion of Participants Requiring Vasopressors for Hypotension
Description: Outcome reported as the number of participants in each arm requiring the use of vasopressors for hypotension.
Time Frame: 10 days
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 102 | 100
proportion of participants | 0.106 | 0.198

4. Secondary Outcome: Proportion of Participants Experiencing Acute Kidney Injury
Description: Outcome reported as the number of participants in each arm who experience acute kidney injury as defined by the Kidney Disease Improving Global Outcomes (KDIGO) guidelines:
  Increase in serum creatinine by 0.3mg/dL or more within 48 hours OR Increase in serum creatinine to 1.5 times baseline or more within the last 7 days OR Urine output less than 0.5 mL/kg/h for 6 hours.
Time Frame: 10 days
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 102 | 100
proportion of participants | 0.106 [0.056 to 0.174] | 0.119 [0.065 to 0.191]

5. Secondary Outcome: Oxygen Saturation / Fractional Inhaled Oxygen (S/F)
Description: Oxygen saturation (percent) is measured by pulse oximeter. Fraction of inspired oxygen (FiO2) (unitless) is the volumetric fraction of oxygen to other gases in respiratory support. The S/F ratio is unitless.
Time Frame: 7 days
Measure: Mean (95% Confidence Interval); unit: n/a (ratio)
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 102 | 100
n/a (ratio) | 357.4 [330.3 to 384.5] | 331.5 [302.0 to 361.0]

6. Secondary Outcome: 28-Day Mortality
Description: Outcome reported as the number of participants who have expired at 28 days post enrollment.
Time Frame: 28 days
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 104 | 101
proportion of participants | 0.087 [0.031 to 0.139] | 0.11 [0.047 to 0.169]

7. Secondary Outcome: 90-Day Mortality
Description: Outcome reported as the number of participants who have expired at 90 days post enrollment.
Time Frame: 90 days
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 104 | 101
proportion of participants | 0.106 [0.045 to 0.163] | 0.11 [0.047 to 0.169]

8. Secondary Outcome: ICU Admission
Description: Outcome reported as the number of participants in each arm who require admission to the Intensive Care Unit (ICU).
Time Frame: 10 days
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 102 | 100
proportion of participants | 0.272 [0.192 to 0.363] | 0.36 [0.270 to 0.457]

9. Secondary Outcome: Number of Ventilator-Free Days
Description: Outcome reported as the mean number of days participants in each arm did not require mechanical ventilation during an in-patient hospital admission.
Time Frame: 28 days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 102 | 100
days | 18.4 [16.5 to 20.4] | 18.1 [16.1 to 20.1]

10. Secondary Outcome: Number of Therapeutic Oxygen-Free Days
Description: Outcome reported as the mean number of days participants in each arm did not require therapeutic oxygen usage during an in-patient hospital admission.
Time Frame: 28 days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 102 | 100
days | 24.6 [23.1 to 26.1] | 23.6 [21.8 to 25.3]

11. Secondary Outcome: Number of Vasopressor-Free Days
Description: Outcome reported as the mean number of days participants in each arm did not require vasopressor usage during an in-patient hospital admission.
Time Frame: 10 days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 102 | 100
days | 9.4 [9.1 to 9.8] | 8.7 [8.2 to 9.3]

12. Secondary Outcome: Length of Hospital Stay
Description: Outcome reported as the mean length of in-patient hospital stay (in days) for participants in each arm.
Time Frame: 90 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 104 | 101
days | 5.9 [4.2 to 7.9] | 7.1 [5.2 to 9.1]

13. Secondary Outcome: Disease Severity Rating
Description: Outcome reported as the number of participants in each arm who fall into each of 7 categories. Lower scores indicate greater condition severity. The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen; 6) Not hospitalized, limitation on activities; 7) Not hospitalized, no limitations on activities.
Time Frame: 28 days
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 102 | 100
score | 4.3 [4.0 to 4.6] | 4.2 [3.8 to 4.5]

14. Secondary Outcome: Change in Viral Load by Nasopharyngeal Swab Day 15
Description: Nasopharyngeal swabs will be collected at baseline and day 15. Viral load is measured as number of viral genetic copies per mL.
Time Frame: 15 days
Measure: Mean (95% Confidence Interval); unit: log10 copies/mL
Arm/Group | Placebo | Losartan
Number analyzed (Participants) | 102 | 100
log10 copies/mL | -4.2 [-5.2 to -3.1] | -4.8 [-5.6 to -3.9]

ADVERSE EVENTS:
Time Frame: 15 days
Description: adverse events were assessed and compared by organ system and not by specific adverse event term
Arm/Group | Placebo | Losartan
All-Cause Mortality (participants affected / at risk) | 11/104 | 11/101
Serious Adverse Events (participants affected / at risk) | 30/104 | 36/101
Other Adverse Events (participants affected / at risk) | 90/104 | 101/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=104) | Losartan (N=101)
Cardiovascular (Cardiac disorders) | 6 (6) | 14 (14)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematologic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neurologic (Nervous system disorders) | 1 (1) | 2 (2)
Renal (Renal and urinary disorders) | 2 (2) | 1 (1)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 19 (19)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=104) | Losartan (N=101)
Cardiovascular (Cardiac disorders) | 24 (24) | 26 (26)
Endocrine (Endocrine disorders) | 1 (1) | 2 (2)
Ear, Nose, and Throat (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 3 (3) | 10 (10)
Genitourinary (Renal and urinary disorders) | 1 (1) | 3 (3)
Hematologic (Blood and lymphatic system disorders) | 6 (6) | 9 (9)
Neurologic (Nervous system disorders) | 4 (4) | 4 (4)
Renal (Renal and urinary disorders) | 21 (21) | 20 (20)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 30 (30)
Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT04312009/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT04312009/ICF_001.pdf